CLINICAL TRIAL: NCT03744715
Title: An Open-Label Extension Study to Allow Continued Dosing and/or Follow-up of Patients Who Have Had Previous Exposure to Poziotinib
Brief Title: A Study to Allow Continued Dosing and/or Follow-up of Patients Who Have Had Previous Exposure to Poziotinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons, not related to safety.
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-POZ-501; 2020-005213-40 (EudraCT Number)
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: NSCLC; Breast Cancer
Keywords: EGFR; HER2; Exon 20 insertion mutation; Poziotinib
MeSH Terms: conditions — Breast Neoplasms | interventions — HM781-36B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Poziotinib (Experimental): Poziotinib will be taken by the patient orally, once daily with food and a glass of water at approximately the same time. The dose will be the last dose received or at the standard starting dose of 16 mg poziotinib. If a dose is missed, it may be taken any time during the day preferably with food, but at least 8 hours prior to the next scheduled dose.
  Interventions: Drug: Poziotinib

INTERVENTIONS:
Drug: Poziotinib — Poziotinib

SUMMARY:
This is an open-label extension study (Extension Study) designed to allow patients to continue to receive poziotinib treatment who have had previous exposure to poziotinib and/or are still receiving clinical benefit from treatment, as judged by the Investigator or treating physician. Patients must begin treatment in this study within 28 days after their last dose of poziotinib.

This extension protocol is intended to provide clinical benefit of poziotinib to patients who are responding to treatment. The additional treatment is optional and voluntary.

DETAILED DESCRIPTION:
Patients who wish to participate in the extension study must provide written Informed Consent. Treatment will begin after completion of the End of Study (EOS) or End of Treatment (EOT) visit of the Original Study. The assessments obtained at the EOS or EOT visit will serve as Baseline data for the extension study.

Patients will continue to receive poziotinib treatment at the last dose received or at the standard starting dose of 16 milligrams (mg) poziotinib, once daily.

Patients may receive treatment as long as the patient is deriving clinical benefit, as judged by the investigator or treating physician (case-by-case decision with approval of Spectrum), death, withdrawal of consent, unacceptable toxicity, lost to follow-up, or poziotinib receives commercial approval in their country of residence or development is terminated by the Sponsor, whichever occurs first. There will be an EOS Visit 35 (±5) days after the last dose of poziotinib.

ELIGIBILITY:
Inclusion Criteria:

* Patient has had previous exposure to poziotinib and is still receiving clinical benefit from treatment, as judged by the Investigator or treating physician.
* Patient must have completed the End of Treatment or End of Study visit if enrolled in a previous (original) poziotinib study.
* Investigator or treating physician opinion indicates that extended therapy with poziotinib is clinically appropriate for the patient and the patient is suitable for this Study.
* Patient agrees to continue study treatment.
* Patient must provide written Informed Consent, must be able to adhere to dosing and visit schedules, and meet protocol-defined study requirements.
* Patient is willing to practice 2 forms of contraception, one of which must be a barrier method, from study entry until at least 30 days after the last dose of poziotinib.

Exclusion Criteria:

* Patient has any ongoing adverse event that hasn't improved to Grade ≤1 and could impact the patient's tolerability to poziotinib.
* Patient has an active uncontrolled infection, bleeding disorder, underlying medical condition, or other serious illness that would impair the ability of the patient to receive poziotinib.
* Patient has any medical or non-medical condition that may not be suitable for poziotinib treatment, as determined by the investigator or treating physician.
* Patient last dose of poziotinib was more than 28 days prior to Day 1 of the study.
* Patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with serious adverse events | 24 months
  Number of patients with serious adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pacific Shores Medical Group, Long Beach, California
  - Hattiesburg Clinic Hematology Oncology, Hattiesburg, Mississippi
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - UPMC, Pittsburgh, Pennsylvania
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided